CLINICAL TRIAL: NCT03033264
Title: A Comparison Between Labor Induction With Dinoprostone and a Cervical Ripening Balloon in Women With a BMI>30 as Oppose With a BMI<30.
Brief Title: Labor Induction With Dinoprostone in Oppose to Cervical Ripening Balloon as a Factor of BMI.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0192-19-RMB
Record Dates: First submitted 2016-12-24; First posted 2017-01-26 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Induction of Labor
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BMI>30+Dinoprostone (Experimental): Women with a BMI>30 at term that will be induced for obstetrical indications with 10 mg of a Dinoprostone vaginal insert.
  Interventions: Drug: Dinoprostone
- BMI<30+Dinoprostone (Experimental): Women with a BMI<30 at term that will be induced for obstetrical indications with 10 mg of a Dinoprostone vaginal insert.
  Interventions: Drug: Dinoprostone
- BMI>30+Cervical ripening balloon (Experimental): Women with a BMI>30 at term that will be induced for obstetrical indications with a double lumen cervical ripening balloon.
  Interventions: Device: Double lumen cervical ripening balloon.
- BMI<30+Cervical ripening balloon (Experimental): Women with a BMI<30 at term that will be induced for obstetrical indications with a double lumen cervical ripening balloon.
  Interventions: Device: Double lumen cervical ripening balloon.

INTERVENTIONS:
Drug: Dinoprostone — 10 mg of a Dinoprostone vaginal insert.
  Other Names: Prostaglandin E2
  Arms: BMI<30+Dinoprostone; BMI>30+Dinoprostone
Device: Double lumen cervical ripening balloon. — Double lumen cervical ripening balloon.
  Arms: BMI<30+Cervical ripening balloon; BMI>30+Cervical ripening balloon

SUMMARY:
Women with a BMI>30 and women with a BMI<30 will be divided in a randomized controlled manor to 4 groups depending on the mode of labor induction and BMI value:

1. Dinoprostone in women with a BMI>30.
2. Dinoprostone in women with a BMI<30.
3. Cervical ripening balloon in women with a BMI>30.
4. Cervical ripening balloon in women with a BMI<30. The subjects will be followed until labor, and information regarding the success of induction, mode of delivery and time of delivery will be collected from patients' electronic files.

DETAILED DESCRIPTION:
The study is a randomized controlled test in which women with a BMI>30 and women with a BMI<30 will sign an informed consent and then divided to 4 groups depending on the mode of labor induction and BMI value:

1. Dinoprostone in women with a BMI>30.
2. Dinoprostone in women with a BMI<30.
3. Cervical ripening balloon in women with a BMI>30.
4. Cervical ripening balloon in women with a BMI<30. All subjects participating in the study will be induced for obstetrical indications alone.

The subjects will be followed until labor, and information regarding the success of induction, mode of delivery and time of delivery will be collected from patients' electronic files.

The participants will finish participation in the study after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant woman at term with an obstetric indication for labor induction.

Exclusion Criteria:

* Previous cesarean section.
* Positive Oxytocin challenge test.
* Positive contraction stress test.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Mode of delivery | Up to 5 days.
  Vaginal delivery in oppose to cesarean section.

SECONDARY OUTCOMES:
Time to delivery | Up to 5 days.
  Time from insertion of induction device\drug until delivery.
Induction success. | Up to 5 days.
  Cervical dilatation and effacement after cessation of induction.
Neonatal complications and outcome. | Up to 5 days.
  Any neonatal complications as mentioned In the neonate's electronic file.

CONTACTS AND LOCATIONS:
Overall Officials: ROY LAUTERBACH, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264